CLINICAL TRIAL: NCT00942201
Title: Comparison of Single Dose Versus Two Doses of Oral Dexamethasone in the Management of Acute Asthma Exacerbations in the Pediatric Emergency Department.
Brief Title: Comparison of Oral Dexamethasone Doses in Asthma Exacerbation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rady Children's Hospital, San Diego (Other)
Responsible Party: Nazli Ghafouri, MD, UC San DIego/Rady Children's Pediatric Emergency Medicine Fellowship
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 080453
Record Dates: First submitted 2009-06-08; First posted 2009-07-20 (Estimated); Last update posted 2009-07-20 (Estimated); Status verified 2009-07

CONDITIONS: Asthma; Reactive Airway Disease
Keywords: Asthma; Dexamethasone; Emergency Department
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Emergencies | interventions — Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single dose dexamethasone (Active Comparator): Single dose dexamethasone 0.6 mg/kg, rounded to nearest 2 mg, max 16 mg administered in ED
  Interventions: Drug: Dexamethasone
- Two dose dexamethasone (Active Comparator): First dose in ED, a prescription for second dose to be administered on Day 3 after discharge
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Single loading dose in ED 0.6 mg/kg, rounded to nearest 2 mg,use 4 mg tabs max dose 16 mg.
  Other Names: Decadron
  Arms: Single dose dexamethasone
Drug: Dexamethasone — Firstdose in ED 0.6 mg/kg, rounded to nearest 2 mg, use 4 mg tabs max dose 16 mg; a prescription for second dose as above to be taken on day 3 after discharge
  Other Names: Decadron
  Arms: Two dose dexamethasone

SUMMARY:
Hypothesis: A 2-day course of oral dexamethasone is the superior option for the resolution of symptoms and prevention of relapse in the emergency department (ED) management of mild-moderate asthma exacerbations.

DETAILED DESCRIPTION:
Asthma has become a major public health problem of increasing concern in the US as it is the most prevalent chronic disease of childhood with over 6 million children under the age of 17 affected 7. Low-income populations, minorities, and children living in inner cities experience disproportionately higher morbidity and mortality due to asthma. Children who suffer from asthma often present to the ED or outpatient center for management of their symptoms and exacerbations. Asthma related ED visits in 2004 were estimated at 1.8 million, with children younger than 17 accounting for almost half with 754,000 visits 7 Recent clinical trials have shown the efficacy of dexamethasone in the ED management of asthma. In Quereshi et al, a randomized study of 533 patients showed that two doses of DEX taken on days 1 and 2 were equally efficacious as 5 days of prednisolone2. However, patients treated with DEX demonstrated improved compliance with less vomiting, fewer missed days of school and fewer missed parental workdays. A more recent study by Altamimi et al compared single dose DEX to 5-day prednisolone1. This double blinded, randomized prospective study of 134 children concluded that single dose DEX is no worse than 5 days of prednisolone as well.dexamethasone in the acute management of asthma exacerbation. However, practices vary as to the use of single dose, two-day dosing and when to administer the second dose. The purpose of this study is to compare various dosing regimes of dexamethasone in its efficacy in the treatment of asthma exacerbations. Given the longer duration of action of DEX (36-72 hours), we hypothesize that 2 doses of DEX given on days 1 & 3 are superior to single dose DEX in improving symptoms and preventing relapse in the ED management of mild to moderate asthma exacerbations.

These previous studies show similar efficacy of dexamethasone when compared to the standard 5-day prednisone/prednisolone treatment. . Within the institution, the investigators have incorporated the use of dexamethasone in the management of acute asthma exacerbations. However, practices vary as to the use of a single dose, two-day dosing and the timing of the second dose for those patients receiving two doses of dexamethasone.

The purpose of this study was to determine if single dose oral dexamethasone is as effective as a 2 dose course of oral dexamethasone in preventing relapse within 7 days for pediatric asthma patients managed in the ED. Given the long half life of dexamethasone, the investigators hypothesized that 2 doses given on days 1 and 3 are superior to single dose in improving symptoms and preventing relapse in the ED management of mild to moderate asthma exacerbations.

ELIGIBILITY:
Inclusion Criteria:

* children 2-17 years old
* with a history of wheezing (> 1 episode requiring ß-2 agonist therapy) who present to the ED with mild to moderate asthma exacerbations

  *mild-moderate exacerbations are defined as a RSS < 11
* patients whose symptoms do not resolve after the first albuterol/atrovent treatment (given in the ED, or at home or via EMS within 1 hour prior to arrival to the ED) are eligible for enrollment

Exclusion Criteria:

* age < 2 years due to overlap with bronchiolitis
* use of steroids within 3 weeks
* recent exposure to TB, varicella, or herpes
* active varicella/herpes infections
* concomitant stridor, vomited 2 doses in ED
* severe asthma as defined by RSS > 12
* requirement for or pre-existing IV access
* need for immediate airway protection
* history of intubations for asthma or comorbidities (Chronic Lung Disease (CLD), Congenital Heart Defects (CHD), or neurologic disorders)

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 125 (Actual)
Dates: Start 2008-08; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
The primary outcome measures are the rate of relapse (including admission to hospital after ED discharge, or unscheduled PCP or ED visits, or new oral corticosteroid prescribed) and time (days) to resolution of symptoms. | Phone follow up on day 7-10 after discharge, day of discharge = day 1. Total duration of study is 10 months.

SECONDARY OUTCOMES:
The secondary outcome measures include compliance, patient/parent satisfaction and rate of hospitalization from the ED. | Phone follow up on day 7-10 after discharge, day of discharge = day 1. Total duration of study is 10 months.

CONTACTS AND LOCATIONS:
Overall Officials: Ghazala Sharieff, MD, Principal Investigator — Rady Children's Hospital
Locations (1):
- Rady Children's Hospital, San Diego, California, United States

REFERENCES:
- [Result] Altamimi S, Robertson G, Jastaniah W, Davey A, Dehghani N, Chen R, Leung K, Colbourne M. Single-dose oral dexamethasone in the emergency management of children with exacerbations of mild to moderate asthma. Pediatr Emerg Care. 2006 Dec;22(12):786-93. doi: 10.1097/01.pec.0000248683.09895.08. PMID 17198210
- [Result] Qureshi F, Zaritsky A, Poirier MP. Comparative efficacy of oral dexamethasone versus oral prednisone in acute pediatric asthma. J Pediatr. 2001 Jul;139(1):20-6. doi: 10.1067/mpd.2001.115021. PMID 11445789
- [Result] Gries DM, Moffitt DR, Pulos E, Carter ER. A single dose of intramuscularly administered dexamethasone acetate is as effective as oral prednisone to treat asthma exacerbations in young children. J Pediatr. 2000 Mar;136(3):298-303. doi: 10.1067/mpd.2000.103353. PMID 10700684
- [Result] Greenberg RA, Kerby G, Roosevelt GE. A comparison of oral dexamethasone with oral prednisone in pediatric asthma exacerbations treated in the emergency department. Clin Pediatr (Phila). 2008 Oct;47(8):817-23. doi: 10.1177/0009922808316988. Epub 2008 May 8. PMID 18467673